CLINICAL TRIAL: NCT04136899
Title: Burn Out and Quality of Life at French General Practioners: is There a Link
Brief Title: Burn Out and Quality of Life at French General Practioners
Status: Completed | Type: Observational
Sponsor: Albert TRINH-DUC (Other)
Responsible Party: Sponsor-Investigator, Albert TRINH-DUC, Thesis Director, Centre Hospitalier St Esprit
Organization: Centre Hospitalier St Esprit (Other)
Other Study IDs: CHSEsprit AGEN
Record Dates: First submitted 2019-08-30; First posted 2019-10-23 (Actual); Last update posted 2019-10-23 (Actual); Status verified 2019-10

CONDITIONS: Cross-Sectional Studies
Keywords: burn out; quality of life; general practioners; french
MeSH Terms: conditions — Burnout, Psychological

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Dukes scale — collection of questionnaires
  Other Names: Maslach Burn-out Inventory Scale

SUMMARY:
The suffering of caregivers is constantly increasing. General medicine, because of its primary role in primary care, is particularly exposed to the risk of burn-out and must protect itself. The aim of this study was to find an inverse relationship between health-related quality of life and being severely burned by French general practitioners.

DETAILED DESCRIPTION:
descriptive quantitative cross-sectional study

ELIGIBILITY:
Inclusion Criteria:

* french general practitioner in liberal activity

Exclusion Criteria:

* retired doctor
* junior general practioner

Ages: 30 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All french general practitioner in activity
Sampling Method: Probability Sample
Enrollment: 1100 (Actual)
Dates: Start 2019-08-20 (Actual); Primary Completion 2019-08-20 (Actual); Study Completion 2019-08-20 (Actual)

PRIMARY OUTCOMES:
Assesment of Burn-out | 30 days
  Maslach Burn-out Inventory scale, 22 Items sort to 0 (never) at 6 (every day) 3 class : An emotional exhaustion (EE), depersonalization (DP) and a reduction of personal accomplishment (AP)
  * The emotional exhaustion (when emotional resources are exhausted, when the workers can no longer give their best, psychologically speaking.)
  * The Depersonalization (reflects withdrawal, indifference to work)
  * The lose of personal accomplishment (devaluation, negative self-evaluation at work)
  Our study focused on severe burn-out, defined by the combination of high EE and DP scores and low AP scores:
  * A high EE is defined by a score > 30
  * A high PD is defined by a score > 12
  * A low PA is defined by a score < 33.
Assesment quality of life: Dukes Scale | 30 days
  The Duke Health Profile 17 items questionnaire. It assesses health-related quality of life and has 10 dimensions.
  The score of each of the 10 dimensions matches with the sum of the item scores, standardized from 0 to 100:
  * For the 6 health scores (general, physical, mental, social, perceived health and self-esteem) 100 specifies the best HRQoL,
  * For the 4 scores of the dysfunction dimension (anxiety, depression, pain, disability), 100 specifies the most significant dysfunction

SECONDARY OUTCOMES:
Socio-demographic data | 30 days
  * age, (years)
  * sex, (female, male)
  * children, (children number)
Mode of practice | 30 days
  * mode of practice (alone, group, liberal..),
  * the number of hours worked, (hours)
  * the number of monthly guards, (months)
  * the number of daily acts, (acts number)
  * the number of weeks of annual leave, (weeks)
Leisure time | 30 days
  * he practice of a sports or leisure activity, (yes, not)
  * he presence or absence of a work stoppage during the last twelve months (weeks)
  * the duration, the need to have had to adjust his working time (yes, not)

CONTACTS AND LOCATIONS:
Overall Officials: Albert TRINH-DUC, MD, Study Director — Centre Hospitalier St Esprit
Locations (1):
- Centre Hospitalier St ESPRIT, Agen, France

IPD SHARING:
Plan to Share IPD: No